CLINICAL TRIAL: NCT02056938
Title: Prospective Multicentric, Randomized, Open-labeled, in Parallel Groups, Study to Assess the Benefit/Risk of an Induction Treatment With Anti-Thymocyte Globulins (ATG) Versus Basiliximab in Kidney Transplant Patients Displaying Low Immunological Risk But High Susceptibility to Delayed Graft Function.
Brief Title: ATG Versus Basiliximab in Kidney Transplant Displaying Low Immunological Risk But High Susceptibility to DGF
Acronym: PREDICT-DGF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment issues
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC14_0051
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Kidney Transplantation
Keywords: Transplantation; kidney; delayed graft function; induction therapy; personalized medicine; First kidney transplantation; No anti HLA immunization prior transplantation; Risk of DGF higher than 40% calculated byt he score DGFS
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATG (Experimental): The first infusion of Thymoglobuline® begins before the kidney reperfusion. In case of a patient with a functional arteriovenous fistula or a high-flow venous catheter, the infusion of Thymoglobuline® can begin just after the randomization pre operatively. When the patient has no available arteriovenous fistula for the Thymoglobuline® infusion, it is necessary to install a high-flow vein (central vein) by the anesthesiologist, and to begin the perfusion as soon as possible intra-operatively before the reperfusion of the kidney. The dose of Thymoglobuline® per infusion is 1.5mg/kg. The duration of each infusion is between 6 to 24 hours.
  The total duration of the Thymoglobuline® administration is 4 days (starting at and including the first day of the surgery).
  Interventions: Drug: Anti-Thymocyte Globulins treatment
- Basiliximab (Active Comparator): The first infusion of Simulect® begins within the two hours before the surgery. There is no need of central venous catheter or arteriovenous fistula to infuse the Simulect®. The duration of the infusion is 30 minutes. Each dose of Simulect® is 20 mg. The first infusion of Simulect® is displayed on Day 0 (within the two hours before the surgery) and the second infusion 3 days afterward (Day 4).
  Interventions: Drug: Basiliximab treatment

INTERVENTIONS:
Drug: Anti-Thymocyte Globulins treatment
  Arms: ATG
Drug: Basiliximab treatment
  Arms: Basiliximab

SUMMARY:
The primary objective of the following randomized open label trial is to demonstrate how low immunological risk patients (no anti HLA immunization and first kidney transplantation) but diagnosed at high-risk of delayed graft function (assessed by DGFS score) could benefit from induction with ATG for preventing delayed graft function compared to Basiliximab.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* First kidney transplantation
* No anti HLA immunization prior transplantation
* A risk of DGF higher than 40% calculated by the score DGFS (DGFS >= 0.4)
* Written informed consent

Exclusion Criteria:

* Previous or combined other transplantations
* Non heart beating donors
* Living donors
* Pre-emptive transplantation
* Patients on peritoneal dialysis
* Leucopenia lower than 3000/mm3
* Thrombopenia lower than 100 000/mm3
* Donor EBV positive / recipient EBV Negative
* Pregnant or lactating women
* Patients under guardianship
* Previous and current history of cancer and/or lymphoma
* Current history of HCV or HBV or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of a delayed graft function | 7 days
  Occurrence of a delayed graft function defined as the need for dialysis within the first seven days post transplantation.

SECONDARY OUTCOMES:
Duration of the delayed graft function | 7 days
  Duration of the DGF defined by the number of days after the transplantation to reach an estimated glomerular filtration rate (eGFR) above 10 mL/min. Only eGFR assessments at least 48 hours after the last day of dialysis will be considered.
Evolution of estimated glomerular filtration rate (eGFR) | 15 days
  Evolution of eGFR from day 1 to day 7 post transplantation then every two days until hospital discharge. Only eGFR assessments at least 48 hours after the last day of dialysis will be considered.
Number of dialysis procedures performed after transplantation without taking into account the dialysis due to hyperkaliemia and/or hyperhydratation | 3 months
Evolution of Tacrolimus levels (T0) from Day 1 to Day 7 post transplantation then every 2 days until hospital discharge. | 15 days
Hematologic effect within the first 3 months of surgery (WBC monitoring, CD3, CD4, CD8, CD19, NK and platelet sub population analysis). | 3 months
Occurrence of infections within the first 3 months post transplantation, especially the CMV and BK reactivation assessed by RTPCR | 3 months
Occurrence of biopsy-confirmed acute rejection episodes and subclinical acute rejection episodes within the first 3 months post transplantation. | 3 months
Percentage of renal fibrosis on a surveillance kidney biopsy at 3 months post transplantation | 3 months
  Percentage of renal fibrosis on a surveillance kidney biopsy at 3 months post transplantation will be evaluated by computerized quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Magali GIRAL, Professor, Principal Investigator — Nantes universitary hospital
Locations (4):
- France (4):
  - Universitary hospital of Lyon, Lyon
  - Nantes Universitary hospital, Nantes
  - Universitary hospital of Nice, Nice
  - Necker Hospital, Paris

REFERENCES:
- [Derived] Chapal M, Foucher Y, Marguerite M, Neau K, Papuchon E, Daguin P, Morelon E, Mourad G, Cassuto E, Ladriere M, Legendre C, Giral M. PREventing Delayed Graft Function by Driving Immunosuppressive InduCtion Treatment (PREDICT-DGF): study protocol for a randomized controlled trial. Trials. 2015 Jun 23;16:282. doi: 10.1186/s13063-015-0807-x. PMID 26099226